CLINICAL TRIAL: NCT03116035
Title: A Randomized Controlled Trial Evaluating the Impact of Pre-Operative Web-based Breast Cancer Information on the Quality of Patient Decision-Making
Brief Title: Impact of Pre-Operative Web-based Breast Cancer Information on the Quality of Patient Decision-Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-1500; UW13089 (Other: UWCCC)
Record Dates: First submitted 2017-04-03; First posted 2017-04-14 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer; Knowledge, Attitudes, Practice
MeSH Terms: conditions — Breast Neoplasms; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based decision aid (Active Comparator): A commercially available web-based breast cancer surgery decision aid
  Interventions: Other: Web-based decision aid
- Standard websites (Active Comparator): selected, high-quality standard web-sites
  Interventions: Other: Standard websites

INTERVENTIONS:
Other: Web-based decision aid — Patients were randomized to receive links to a commercially available decision aid.
  Arms: Web-based decision aid
Other: Standard websites — Patients were randomized to receive links to standard, high-quality websites.
  Arms: Standard websites

SUMMARY:
This is a prospective randomized control trial to compare the impact of two different types of pre-operative web-based breast cancer information on the quality of patient decision making. Patients are emailed web-based information prior to the surgical consultation. Outcomes are assess at multiple time points: 1) prior to the surgical consultation, 2) immediately following the consultation.

ELIGIBILITY:
1. >18 years of age
2. Newly diagnosed stage 0-3 breast cancer
3. English speaking
4. Has an email address
5. No prior recent contact with the breast surgeon

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2014-04-24 (Actual); Primary Completion 2016-06-28 (Actual); Study Completion 2016-06-28 (Actual)

PRIMARY OUTCOMES:
Knowledge using the Breast Cancer Decision Quality Instrument | immediately prior to the surgical consultation

SECONDARY OUTCOMES:
Decisional concordance using the Breast Cancer Decision Quality Instrument | immediately prior to the surgical consultation
Perceived communication with the breast surgeon using the Breast Cancer Decision Quality Instrument | following the surgical consultation but prior to the surgery
Breast surgeon and staff (nurse, mid-level provider) assessment of how the web-based decision aid versus standard high-quality breast cancer websites influenced their patient interactions, based on Practitioner Opinion Survey | at completion of patient accrual, estimated to be 2 years after initiating study

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tucholka JL, Yang DY, Bruce JG, Steffens NM, Schumacher JR, Greenberg CC, Wilke LG, Steiman J, Neuman HB. A Randomized Controlled Trial Evaluating the Impact of Web-Based Information on Breast Cancer Patients' Knowledge of Surgical Treatment Options. J Am Coll Surg. 2018 Feb;226(2):126-133. doi: 10.1016/j.jamcollsurg.2017.10.024. Epub 2017 Dec 12. PMID 29246705